CLINICAL TRIAL: NCT02104076
Title: Evaluation for the Effectiveness of Evolution® Biliary Stent System-Fully Covered
Brief Title: Evolution® Biliary Stent System-Fully Covered
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 10-014
Record Dates: First submitted 2014-04-02; First posted 2014-04-04 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-06

CONDITIONS: Carcinomas/Neoplasms
Keywords: Bile Duct Obstructions; Biliary Stases; Biliary Tract; Stents
MeSH Terms: conditions — Carcinoma; Neoplasms; Cholestasis

ARMS (1):
- Evolution® Biliary Stent-Fully Covered (Experimental)
  Interventions: Device: Evolution® Biliary Stent-Fully Covered

INTERVENTIONS:
Device: Evolution® Biliary Stent-Fully Covered — Implantation of the Evolution® Biliary Stent-Fully Covered in the common bile duct utilizing ERCP

SUMMARY:
The Evolution® Biliary Stent System-Fully Covered study is a clinical trial approved by the US FDA to evaluate the effectiveness of the Evolution® Biliary Stent System-Fully Covered when used in palliation of malignant neoplasms in the biliary tree.

ELIGIBILITY:
Inclusion Criteria:

* Inoperable malignant neoplasm causing biliary obstruction or stricture that requires a fully covered metal stent

Exclusion Criteria:

* < 18 years of age
* Unwilling or unable to sign and date the informed consent
* Unwilling or unable to comply with the follow-up schedule
* Undergone or is planning to undergo brachytherapy with transpapillary or percutaneous implantation of intracavitary radiation sources
* Participating in another investigational drug or device study in which patient has not completed the follow-up phase for the primary endpoint at least 30 days prior to enrollment
* Endoscopic procedures are contraindicated
* Current anatomy upstream of intended stent placement compromising the flow of bile from the liver such that stent placement may not alleviate the biliary obstruction symptoms
* Presence of a metal biliary stent
* Presence of an esophageal or duodenal stent
* Hypersensitivity/allergy or contraindication to any component of the stent, delivery system, or medication required to complete the procedure,which in the investigator's opinion cannot be adequately premedicated
* Coagulopathy
* Diffuse intrahepatic metastases that involves > 10 % of the liver
* Life expectancy of < 3 months
* Pregnant
* Active alcohol or substance abuse issue
* Jaundice secondary to a cause other than biliary duct obstruction
* Additional endoscopic restrictions as specified in the Clinical Investigation Plan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-09; Primary Completion 2016-07 (Actual); Study Completion 2017-01-04 (Actual)

PRIMARY OUTCOMES:
Percentage of patients free from symptomatic recurrent of biliary obstruction requiring reintervention | 6 months
Total Serum Bilirubin ≤ 3.0 mg/dL | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Raj Shah, M.D., Principal Investigator — University of Colorado, Denver; Marco Bruno, M.D., Principal Investigator — Erasmus Medish Centrum
Locations (12):
- United States (7):
  - University of Colorado Hospital, Aurora, Colorado
  - Borland-Groover Clinic, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Indiana University Hospital, Indianapolis, Indiana
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Virginia Health System, Charlottesville, Virginia
- Canada (2):
  - St. Michael's Hospital, Toronto, Ontario
  - Centre Hospitalier de 1'Université, Montreal, Quebec
- France (2):
  - Hôpital Edouard Herriot, Lyon
  - Hôpital L'Archet 2, Nice
- Erasmus Medish Centrum, Rotterdam, Netherlands